CLINICAL TRIAL: NCT01646073
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Assess the Safety and Efficacy of Adalimumab (Humira®) in Chinese Subjects With Moderate to Severe Plaque Psoriasis
Brief Title: Safety and Efficacy Study of Adalimumab in the Treatment of Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M13-606
Record Dates: First submitted 2012-07-18; First posted 2012-07-20 (Estimated); Results first posted 2015-01-19 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2015-01

CONDITIONS: Plaque Psoriasis
Keywords: Plaque Psoriasis; Psoriasis; Placebo Controlled; Skin Disease; Double Blind
MeSH Terms: conditions — Psoriasis; Skin Diseases | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adalimumab (Experimental): Adalimumab 40 mg every other week (eow)
  Interventions: Biological: Adalimumab
- Placebo (Placebo Comparator): placebo
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: Adalimumab — adalimumab eow
  Other Names: ABT-D2E7; Humira
  Arms: Adalimumab
Biological: placebo — placebo
  Arms: Placebo

SUMMARY:
A study to evaluate the safety and efficacy of adalimumab in Chinese subjects with moderate to severe plaque psoriasis.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and efficacy of adalimumab and to determine how well it works in the treatment of adults with moderate to severe plaque psoriasis in the Chinese population. Psoriasis is a chronic immunologic disease characterized by marked inflammation and thickening of the epidermis that result in thick, scaly plaques involving the skin.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of psoriasis for at least 6 months.
* Must have stable plaque psoriasis for at least 2 months before screening and baseline visits.
* Participant must have a Psoriasis Area Severity Index score greater than or equal to 10 at the baseline visit.
* Participant must have moderate to severe plaque Psoriasis, defined by Body Surface Area involvement greater than or equal to 10% at the baseline visit.
* Participant must have a Physicians Global Assessment of at least moderate disease at baseline visit.

Exclusion Criteria:

* Diagnosis of other active skin diseases or skin infections.
* Participant has known hypersensitivity to adalimumab or it excipients.
* Participant has chronic recurring infections or active tuberculosis.
* Participant has demyelinating disease (including myelitis) or neurologic symptoms suggestive of demyelinating disease.
* Participant is known to have immune deficiency or is immunocompromised.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 425 (Actual)
Dates: Start 2012-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Okun, MD, Study Chair — AbbVie
Locations (16):
- China (16):
  - Site Reference ID/Investigator# 72888, Beijing
  - Site Reference ID/Investigator# 72873, Beijing
  - Site Reference ID/Investigator# 72887, Beijing
  - Site Reference ID/Investigator# 85693, Chengdu
  - Site Reference ID/Investigator# 72976, Chongqing
  - Site Reference ID/Investigator# 72880, Dalian
  - Site Reference ID/Investigator# 72973, Guangzhou
  - Site Reference ID/Investigator# 72974, Guangzhou
  - Site Reference ID/Investigator# 72878, Hangzhou, Zhejiang
  - Site Reference ID/Investigator# 72877, Hangzhou, Zhejiang
  - Site Reference ID/Investigator# 87058, Jinan
  - Site Reference ID/Investigator# 72876, Shanghai
  - Site Reference ID/Investigator# 72875, Shanghai
  - Site Reference ID/Investigator# 72883, Shenyang
  - Site Reference ID/Investigator# 72977, Wuhan, Hubei
  - Site Reference ID/Investigator# 72975, Xi'an

REFERENCES:
- See also: Related Info — http://www.rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized at Week 0 (Day 1) in a 4:1 ratio to receive either adalimumab every other week (eow) or matching placebo.
Groups:
- Placebo: Participants were started on placebo in Period A and then switched to adalimumab 40 mg eow in Period B
- Adalimumab Eow: Participants were started on 40 mg adalimumab every other week (eow) in Period A and continued adalimumab 40 mg eow into Period B
Period: Period A (12 Weeks)
Arm/Group | Placebo | Adalimumab Eow
Started | 87 | 338
Completed | 85 | 333
Not Completed | 2 | 5
Not completed — Adverse Event | 0 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Other | 0 | 1
Period: Period B (12 Weeks)
Arm/Group | Placebo | Adalimumab Eow
Started | 85 | 333
Completed | 84 | 320
Not Completed | 1 | 13
Not completed — Adverse Event | 0 | 7
Not completed — Withdrawal by Subject | 1 | 5
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants were started on placebo in Period A and then switched to 40 mg adalimumab eow in Period B
- Adalimumab Eow: Participants were started on adalimumab 40 mg every other week (eow) in Period A and continued adalimumab 40 mg eow into Period B
- Total: Total of all reporting groups
Arm/Group | Placebo | Adalimumab Eow | Total
Number analyzed (Participants) | 87 | 338 | 425
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (12.45) | 43.1 (11.91) | 43.2 (12.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 84 | 113
  Male | 58 | 254 | 312
Duration of Psoriasis [Mean (Standard Deviation); unit: years] | 15.79 (10.309) | 14.84 (10.114) | 15.03 (10.149)
Body Surface Area with Psoriasis [Mean (Standard Deviation); unit: Percentage of Body Surface Area] | 39.30 (22.502) | 42.62 (21.748) | 41.94 (21.918)
Psoriasis Area and Severity Index [Mean (Standard Deviation); unit: units on a scale] — Psoriasis Area and Severity Index (PASI) is a composite measure of the level of erythema (redness of the skin), induration (hardening of the skin), and desquamation (peeling of the skin) on 4 sites (head, upper extremities, trunk, and lower extremities), each of which are rated on a 5-point scale from 0 (no symptoms) to 4 (very marked). The possible range for PASI score is 0 to 72, with the highest score representing complete erythroderma of the severest possible degree; a decrease in score indicates improvement.
  units on a scale | 25.60 (10.978) | 28.19 (11.999) | 27.66 (11.831)
Physician's Global Assessment of Psoriasis [Number; unit: participants]
  Clear | 0 | 0 | 0
  Minimal | 0 | 0 | 0
  Mild | 0 | 0 | 0
  Moderate | 57 | 214 | 271
  Marked | 28 | 110 | 138
  Severe | 2 | 14 | 16

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving a Psoriasis Area and Severity Index Greater Than or Equal to 75% Reduction (PASI 75) Response at Week 12
Description: The percentage of participants with a greater than or equal to 75% reduction (improvement) in Psoriasis Area and Severity Index (PASI) score at Week 12. PASI is a composite measure of the level of erythema (redness of the skin), induration (hardening of the skin), and desquamation (peeling of the skin) on 4 sites (head, upper extremities, trunk, and lower extremities), each of which are rated on a 5-point scale from 0 (no symptoms) to 4 (very marked). The possible range for PASI score is 0 to 72, with the highest score representing complete erythroderma of the severest possible degree; a decrease in score indicates improvement.
Time Frame: Week 12
Population: Intent to Treat Population A (ITT_A): all participants who were randomized at Week 0 (Baseline); Non-responder imputation (NRI): any participant who had a missing value at a specific visit as non-responder for that visit.
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Participants were started on placebo in Period A (Week 0 to Week 12).
- Adalimumab Eow: Participants were started on 40 mg adalimumab eow in Period A (Week 0 to Week 12).
Arm/Group | Placebo | Adalimumab Eow
Number analyzed (Participants) | 87 | 338
percentage of participants | 11.5 | 77.8

2. Secondary Outcome: Percentage of Participants Achieving a Psoriasis Area and Severity Index Greater Than or Equal to 75% Reduction (PASI 75) Response [Period A]
Description: The percentage of participants with a greater than or equal to 75% reduction (improvement) in Psoriasis Area and Severity Index (PASI), other than Week 12. PASI is a composite measure of the level of erythema (redness of the skin), induration (hardening of the skin), and desquamation (peeling of the skin) on 4 sites (head, upper extremities, trunk, and lower extremities), each of which are rated on a 5-point scale from 0 (no symptoms) to 4 (very marked). The possible range for PASI score is 0 to 72, with the highest score representing complete erythroderma of the severest possible degree; a decrease in score indicates improvement.
Time Frame: Weeks 3 and 7
Population: ITT_A: all participants that were randomized in Week 0 (Baseline); NRI: any participant who had a missing value at a specific visit as non-responder for that visit.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Adalimumab Eow
Number analyzed (Participants) | 87 | 338
percentage of participants
  Week 3 | 0 | 9.8
  Week 7 | 2.3 | 45.3

3. Secondary Outcome: Percentage of Participants Achieving a Psoriasis Area and Severity Index Greater Than or Equal to 75% Reduction (PASI 75) Response [Period B]
Description: The percentage of participants with a greater than or equal to 75% reduction (improvement) in Psoriasis Area and Severity Index (PASI). PASI is a composite measure of the level of erythema (redness of the skin), induration (hardening of the skin), and desquamation (peeling of the skin) on 4 sites (head, upper extremities, trunk, and lower extremities), each of which are rated on a 5-point scale from 0 (no symptoms) to 4 (very marked). The possible range for PASI score is 0 to 72, with the highest score representing complete erythroderma of the severest possible degree; a decrease in score indicates improvement.
Time Frame: Weeks 16, 19, and 24
Population: Intent to Treat Population B (ITT_B): all participants who received at least 1 dose of study drug in Period B; NRI: any participant who had a missing value at a specific visit as non-responder for that visit.
Measure: Number; unit: percentage of participants
Groups:
- Placebo/Adalimumab Eow: Participants were started on placebo in Period A and then switched to 40 mg adalimumab eow in Period B (Week 12 to Week 24).
- Adalimumab Eow/Adalimumab Eow: Participants were started on 40 mg adalimumab eow in Period A and continued 40 mg adalimumab eow in Period B (Week 12 to Week 24).
Arm/Group | Placebo/Adalimumab Eow | Adalimumab Eow/Adalimumab Eow
Number analyzed (Participants) | 85 | 333
percentage of participants
  Week 16 | 51.8 | 87.4
  Week 19 | 80.0 | 87.1
  Week 24 | 90.6 | 87.7

4. Secondary Outcome: Percent Change From Baseline in Psoriasis Area and Severity Index (PASI) Score [Period A]
Description: Psoriasis Area and Severity Index (PASI), is a composite measure of the level of erythema (redness of the skin), induration (hardening of the skin), and desquamation (peeling of the skin) on 4 sites (head, upper extremities, trunk, and lower extremities), each of which are rated on a 5-point scale from 0 (no symptoms) to 4 (very marked). The possible range for PASI score is 0 to 72, with the highest score representing complete erythroderma of the severest possible degree; a decrease in score indicates improvement.
Time Frame: Baseline to Week 12
Population: ITT_A: all participants that were randomized in Week 0 (Baseline); Last observation carried forward (LOCF): used the completed evaluation from the previous visit within the particular period for efficacy measures assessed to impute missing data at later visits in the same period. Baseline efficacy evaluations were not carried forward.
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Adalimumab Eow
Number analyzed (Participants) | 87 | 336
Percent change | -20.44 (3.049) | -82.20 (1.548)

5. Secondary Outcome: Percent Change From Baseline in Psoriasis Area and Severity Index (PASI) Score [Period B]
Description: PASI is a composite measure of the level of erythema (redness of the skin), induration (hardening of the skin), and desquamation (peeling of the skin) on 4 sites (head, upper extremities, trunk, and lower extremities), each of which are rated on a 5-point scale from 0 (no symptoms) to 4 (very marked). The possible range for PASI score is 0 to 72, with the highest score representing complete erythroderma of the severest possible degree; a decrease in score indicates improvement.
Time Frame: Baseline to Week 24
Population: ITT_B: all participants who received at least 1 dose of study drug in Period B; LOCF: used the completed evaluation from the previous visit within the particular period for efficacy measures assessed to impute missing data at later visits in the same period. Baseline efficacy evaluations were not carried forward.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo/Adalimumab Eow | Adalimumab Eow/Adalimumab Eow
Number analyzed (Participants) | 85 | 333
percent change | -91.39 (14.423) | -91.07 (19.028)

6. Secondary Outcome: Percentage of Participants Achieving a Psoriasis Area and Severity Index Greater Than or Equal to 50%, 90%, or 100% Reduction (PASI 50/90/100) Response [Period A]
Description: The percentage of participants with a greater than or equal to 50%, 90%, or 100% reduction (improvement) in Psoriasis Area and Severity Index (PASI 50/90/100). PASI is a composite measure of the level of erythema (redness of the skin), induration (hardening of the skin), and desquamation (peeling of the skin) on 4 sites (head, upper extremities, trunk, and lower extremities), each of which are rated on a 5-point scale from 0 (no symptoms) to 4 (very marked). The possible range for PASI score is 0 to 72, with the highest score representing complete erythroderma of the severest possible degree; a decrease in score indicates improvement.
Time Frame: Weeks 3, 7, and 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Adalimumab Eow
Number analyzed (Participants) | 87 | 338
percentage of participants
  PASI 50 [Week 3] | 1.1 | 31.7
  PASI 90 [Week 3] | 0 | 2.7
  PASI 100 [Week 3] | 0 | 0
  PASI 50 [Week 7] | 11.5 | 77.2
  PASI 90 [Week 7] | 0 | 23.4
  PASI 100 [Week 7] | 0 | 3.8
  PASI 50 [Week 12] | 23.0 | 88.8
  PASI 90 [Week 12] | 3.4 | 55.6
  PASI 100 [Week 12] | 1.1 | 13.3

7. Secondary Outcome: Percentage of Participants Achieving a Psoriasis Area and Severity Index Greater Than or Equal to 50%, 90%, or 100% Reduction (PASI 50/90/100) Response [Period B]
Description: as for outcome 6
Time Frame: Weeks 16, 19, and 24
Population: ITT_B: all participants who received at least 1 dose of study drug in Period B; NRI: any participant who had a missing value at a specific visit as non-responder for that visit.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo/Adalimumab Eow | Adalimumab Eow/Adalimumab Eow
Number analyzed (Participants) | 85 | 333
percentage of participants
  PASI 50 [Week 16] | 71.8 | 93.4
  PASI 90 [Week 16] | 28.2 | 70.0
  PASI 100 [Week 16] | 8.2 | 20.4
  PASI 50 [Week 19] | 92.9 | 94.3
  PASI 90 [Week 19] | 56.5 | 74.2
  PASI 100 [Week 19] | 22.4 | 28.8
  PASI 50 [Week 24] | 94.1 | 91.9
  PASI 90 [Week 24] | 75.3 | 76.3
  PASI 100 [Week 24] | 34.1 | 35.7

8. Secondary Outcome: Percentage of Participants With a Physician's Global Assessment (PGA) of "Clear" [Period A]
Description: The Physician's Global Assessment (PGA) is a 6-point scale used to measure the severity of disease at the time of the physician's evaluation of the participant ranging from 'clear' (meaning no signs of plaque) to 'severe.'
Time Frame: Baseline and Weeks 3, 7, and 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Adalimumab Eow
Number analyzed (Participants) | 87 | 338
percentage of participants
  Baseline | 0 | 0
  Week 3 | 0 | 0.6
  Week 7 | 0 | 12.1
  Week 12 | 1.1 | 25.7

9. Secondary Outcome: Percentage of Participants With a Physician's Global Assessment (PGA) of "Clear" [Period B]
Description: as for outcome 8
Time Frame: Weeks 16, 19, and 24
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Placebo/Adalimumab Eow | Adalimumab Eow/Adalimumab Eow
Number analyzed (Participants) | 85 | 333
percentage of participants
  Week 16 | 14.1 | 39.3
  Week 19 | 29.4 | 42.9
  Week 24 | 41.2 | 45.6

10. Secondary Outcome: Percentage of Participants With a Physician's Global Assessment (PGA) of "Clear" or "Minimal" [Period A]
Description: as for outcome 8
Time Frame: Baseline and Weeks 3, 7, and 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Adalimumab Eow
Number analyzed (Participants) | 87 | 338
percentage of participants
  Baseline | 0 | 0
  Week 3 | 0 | 20.1
  Week 7 | 4.6 | 57.4
  Week 12 | 14.9 | 80.5

11. Secondary Outcome: Percentage of Participants With a Physician's Global Assessment (PGA) of "Clear" or "Minimal" [Period B]
Description: as for outcome 8
Time Frame: Weeks 16, 19, and 24
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Placebo/Adalimumab Eow | Adalimumab Eow/Adalimumab Eow
Number analyzed (Participants) | 85 | 333
percentage of participants
  Week 16 | 61.2 | 85.6
  Week 19 | 84.7 | 84.4
  Week 24 | 89.4 | 83.8

12. Secondary Outcome: Percentage of Participants Achieving a Dermatology Life Quality Index (DLQI) Score of "0" [Period A]
Description: The DLQI measures how much a subject's skin problem affected their life over the last week. The possible range for DLQI was 0 to 30, with a higher score indicating a more impaired quality of life; a decrease in score indicates improvement.
Time Frame: Baseline, Week 3, and Week 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Adalimumab Eow
Number analyzed (Participants) | 87 | 338
percentage of participants
  Baseline | 0 | 0.9
  Week 3 | 1.1 | 3.3
  Week 12 | 0 | 13.0

13. Secondary Outcome: Percentage of Participants Achieving a Dermatology Life Quality Index (DLQI) Score of "0" [Period B]
Description: The DLQI measures how much a participant's skin problem affected their life over the last week. The possible range for DLQI was 0 to 30, with a higher score indicating a more impaired quality of life; a decrease in score indicates improvement.
Time Frame: Week 16 and Week 24
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Placebo/Adalimumab Eow | Adalimumab Eow/Adalimumab Eow
Number analyzed (Participants) | 85 | 333
percentage of participants
  Week 16 | 12.9 | 15.0
  Week 24 | 23.5 | 19.5

14. Secondary Outcome: Percentage of Participants Achieving a Dermatology Life Quality Index (DLQI) Score of "0 or 1" [Period A]
Description: as for outcome 12
Time Frame: Baseline, Week 3, and Week 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Adalimumab Eow
Number analyzed (Participants) | 87 | 338
percentage of participants
  Baseline | 1.1 | 2.4
  Week 3 | 3.4 | 9.2
  Week 12 | 10.3 | 28.4

15. Secondary Outcome: Percentage of Participants Achieving a Dermatology Life Quality Index (DLQI) Score of "0 or 1" [Period B]
Description: as for outcome 13
Time Frame: Week 16 and Week 24
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Placebo/Adalimumab Eow | Adalimumab Eow/Adalimumab Eow
Number analyzed (Participants) | 85 | 333
percentage of participants
  Week 16 | 27.1 | 30.0
  Week 24 | 44.7 | 37.8

16. Secondary Outcome: Change From Baseline in the Short Form 36 (SF-36) Physical Component Score (PCS) and Mental Component Score (MCS) [Period A]
Description: Short Form-36 is a generic 36-item questionnaire measuring health-related quality of life (HRQL) covering 2 summary measures: physical component summary (PCS) and mental component summary (MCS). The SF-36 consists of 8 subscales. The PCS is represented by 4 subscales: physical function, role limitations due to physical problems, bodily pain, and general health perception. The MCS is represented by 4 subscales: vitality, social function, role limitations due to emotional problems, and mental health. Participants self-report on items in a subscale that have choices per item. Summations of item scores of the same subscale give the subscale scores, which were transformed into a range from 0 to 100; zero= worst HRQL, 100=best HRQL. PCS and MCS scores were constructed as a T-score with a mean of 50 and standard deviation of 10 and no minimum or maximum score. The difference from baseline to week 12 in SF-36 PCS and MCS was calculated.
Time Frame: Baseline to Week 12
Population: ITT_A: all participants that were randomized in Week 0 (Baseline); LOCF: used the completed evaluation from the previous visit within the particular period for efficacy measures assessed to impute missing data at later visits in the same period. Baseline efficacy evaluations were not carried forward.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Adalimumab Eow
Number analyzed (Participants) | 84 | 335
scores on a scale
  Physical Component Summary | 1.13 (0.665) | 4.22 (0.332)
  Mental Component Summary | 1.91 (0.913) | 7.02 (0.456)

17. Secondary Outcome: Change From Baseline in the Short Form 36 (SF-36) Physical Component Score (PCS) and Mental Component Score (MCS) [Period B]
Description: as for outcome 16
Time Frame: Baseline to Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo/Adalimumab Eow | Adalimumab Eow/Adalimumab Eow
Number analyzed (Participants) | 84 | 332
scores on a scale
  Physical Component Summary | 4.20 (8.351) | 4.73 (8.260)
  Mental Component Summary | 5.74 (12.661) | 7.76 (11.652)

ADVERSE EVENTS:
Time Frame: Baseline up to 70 days after last dose (week 24).
Groups:
- Double-blind Placebo: Participants were started on placebo in Period A (Week 0 to Week 12)
- Double-blind Adalimumab Eow: Participants were started on adalimumab eow in Period A (Week 0 to Week 12)
- Any Adalimumab: Participants that received at least one dose of adalimumab during Period A or Period B
Arm/Group | Double-blind Placebo | Double-blind Adalimumab Eow | Any Adalimumab
Serious Adverse Events (participants affected / at risk) | 3/87 | 4/338 | 15/423
Other Adverse Events (participants affected / at risk) | 14/87 | 64/338 | 137/423
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Placebo (N=87) | Double-blind Adalimumab Eow (N=338) | Any Adalimumab (N=423)
ARRHYTHMIA (Cardiac disorders) | 0 | 0 | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 | 0 | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 1 | 1
MYOCARDITIS (Cardiac disorders) | 0 | 0 | 1
PYLORIC STENOSIS (Congenital, familial and genetic disorders) | 0 | 0 | 1
RETINAL DETACHMENT (Eye disorders) | 1 | 0 | 0
GASTRIC ULCER (Gastrointestinal disorders) | 0 | 0 | 1
LUNG INFECTION (Infections and infestations) | 0 | 0 | 2
LYMPH NODE TUBERCULOSIS (Infections and infestations) | 0 | 0 | 1
PNEUMONIA (Infections and infestations) | 0 | 0 | 2
TUBERCULOSIS (Infections and infestations) | 0 | 0 | 1
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 1
SKIN INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 1
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
PSORIATIC ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
ENDOMETRIAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
CEREBRAL INFARCTION (Nervous system disorders) | 0 | 1 | 1
HAEMATURIA (Renal and urinary disorders) | 0 | 1 | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
PLEURAL FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
ERYTHEMA MULTIFORME (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
PSORIASIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
HYPERTENSION (Vascular disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Placebo (N=87) | Double-blind Adalimumab Eow (N=338) | Any Adalimumab (N=423)
NASOPHARYNGITIS (Infections and infestations) | 5 | 13 | 38
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 6 | 34 | 68
COUGH (Respiratory, thoracic and mediastinal disorders) | 4 | 11 | 27
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 14 | 30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.